CLINICAL TRIAL: NCT05907889
Title: FoodSEqual Food Study
Acronym: FOODY
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Reading (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Principal Investigator, Gunter G C Kuhnle, Professor of Nutrition and Health, University of Reading
Other Study IDs: FS_BM_01
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, Hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diet is an important modifiable risk factor for many chronic diseases, but there is a paucity of dietary data from disadvantaged communities. The last Low Income Diet and Nutrition Survey (LIDNS) was conducted more than a decade ago and disadvantaged communities are known to be under-represented in other national surveys.

The aim of the study is to investigate diet and health and factors contributing to dietary choice in a sample of socio-culturally diverse disadvantaged communities using a combination of dietary intake assessment methods, including nutritional biomarkers

DETAILED DESCRIPTION:
The FoodSEqual project is part of a five-year national consortium project led by the University of Reading and involves academics from Plymouth, Sussex, Kent and Cranfield Universities. It is funded by the UK Research and Innovation (UKRI) Strategic Priorities Fund (SPF). The vision of the FoodSEqual project is to provide citizens of socio-culturally diverse disadvantaged communities with choice and agency over the food they consume by co-developing new products, new supply chains and new policy frameworks that deliver affordable, attractive, healthy, and sustainable diet. The FoodSEqual Health project is a follow-on project to investigate associations between diet, health, and food affordability in the context of the FoodSEqual project.

Diet is an important modifiable risk factor for many chronic diseases, but there is a paucity of dietary data from disadvantaged communities. The last Low Income Diet and Nutrition Survey (LIDNS) was conducted more than a decade ago and disadvantaged communities are known to be under-represented in other national surveys.

The aim of the study is to investigate diet and factors contributing to dietary choice in a sample of socio-culturally diverse disadvantaged communities using a combination of dietary intake assessment methods, including nutritional biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over

Exclusion Criteria:

* unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General public
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Food intake | 18 months
  Habitual dietary intake using biomarkers, FFQ and 24h recall

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No